CLINICAL TRIAL: NCT06518005
Title: An Open-label, Phase 2 Trial to Evaluate the Efficacy and Safety of a Single Intravenous Administration of GNT0003 (an Adeno-associated Viral (AAV) Vector Expressing the UGT1A1 Transgene) Following Imlifidase Pre-treatment in Adult Participants With Severe Crigler-Najjar Syndrome (CNS) Requiring Daily Phototherapy and Presenting Pre-existing Anti-AAV8 Antibodies
Brief Title: Efficacy and Safety of GNT0003 Following Imlifidase Pre-treatment in Severe Crigler-Najjar Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genethon (Other)
Collaborators: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNT-018-IDES
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-07

CONDITIONS: Crigler-Najjar Syndrome
MeSH Terms: conditions — Crigler-Najjar Syndrome | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with imlifidase (Experimental): Each participant will be treated with imlifidase
  Interventions: Drug: Imlifidase
- Treatment with GNT0003 (Experimental): Each participant will be treated with GNT0003
  Interventions: Drug: GNT0003

INTERVENTIONS:
Drug: Imlifidase — Imlifidase: single administration (dose is confidential), Lyophilized powder for concentrate for solution for infusion
  Arms: Treatment with imlifidase
Drug: GNT0003 — GNT0003: single administration 5E+12 VG/kg, Sterile concentrate for solution for infusion
  Arms: Treatment with GNT0003

SUMMARY:
Clinical trial rationale:

CNS is an ultra-rare (<1/1 million newborns), autosomal recessive disorder of bilirubin conjugation caused by mutation in the gene coding for uridine 5'-diphosphate glucuronosyltransferase (UGT1A1), that causes the accumulation of neurotoxic unconjugated bilirubin (UCB).

Reduction of UCB is managed with phenobarbital in mild CNS, and daily phototherapy in severe CNS.

There is no authorized curative medical treatment for CNS. Liver transplantation is currently the only curative treatment for severe CNS.

GNT0003 is a genetically modified recombinant (r) viral vector composed of the AAV8 viral capsid carrying the UGT1A1 transgene which aims to correct the dysfunction of the mutated gene by achieving durable expression of a functional copy of the affected gene.

Imlifidase (IgG-degrading enzyme) has demonstrated its efficacy in highly sensitized adult kidney transplant patients.

To give participants with pre-existing anti-AAV8 antibodies access to gene therapy treatments, this trial aims to demonstrate the safety and efficacy of GNT0003 following imlifidase pre-treatment in adult participants with severe CNS requiring daily phototherapy and presenting with pre-existing anti-AAV8 antibodies.

Primary objective: to assess efficacy of a single intravenous administration of GNT0003 following imlifidase pre-treatment in participants with severe CNS requiring phototherapy and pre-existing AAV8 antibodies

Secondary objective: to collect data on safety and tolerability of GNT0003 and imlifidase, efficacy of imlifidase, pharmacokinetic and pharmacodynamic profile of GNT0003, and Quality of Life.

The trial will include 3 parts:

* A baseline period for at least 3 months
* A treatment period
* A follow-up period:

  * Initial post-treatment follow-up over 48 weeks
  * Long-term follow-up for 4 additional years

This trial will be conducted in accordance with the International Conference on Harmonization Guideline for Good Clinical Practice and the Declaration of Helsinki. Participants must be consented using the approved Informed Consent Form before any procedures specified in the protocol are performed.

ELIGIBILITY:
Main Inclusion Criteria:

1. Severe Crigler-Najjar syndrome requiring ≥ 6 hours/ day of phototherapy
2. Molecular confirmation of mutation in the UGT1A1gene by DNA sequencing
3. Detectable serum neutralizing antibodies against AAV8
4. Laboratory parameters value not clinically significant
5. Highly effective method of contraception
6. Affiliated to or a beneficiary of a health care system

Exclusion Criteria:

1. Participation in another interventional trial within 6 months prior to start of clinical trial intervention and during the whole clinical trial
2. Fibrosis score ≥ 3 (METAVIR) or 10 kPa (FibroScan®)
3. Liver transplantation
4. Significant underlying liver disease, chronic hepatitis B, C and/or infected with Human immunodeficiency virus
5. Any other clinically significant illness
6. Uncontrolled hyperlipidemia.
7. History of major thrombotic events, active peripheral vascular disease, proven hypercoagulable conditions,
8. History or presence of thrombotic thrombocytopenic purpura (TTP) or known familial history of TTP
9. Prior or current treatment with Gene therapy, cell based therapy, CRISPR/Cas9 or any other form of gene editing, imlifidase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with serum total bilirubin ≤ 300 μmol/L, 48 weeks after GNT0003 infusion and without phototherapy from Week 16 | 48 weeks post GNT0003 administration
  Decrease of serum total bilirubin level after interruption of daily phototherapy; change in serum total bilirubin from baseline to week 48.

SECONDARY OUTCOMES:
Incidence of significant clinical and/or laboratoy abnormalities, of all treatment-emergent adverse events, serious adverse events, adverse events of special interrests, adverse drug reactions, malignancies | 48 weeks; 60 months
  Incidence and severity for each body system and laboratory parameter will be presented and summarized overall
Change in Health-related quality of Life form baseline to week 48 post GNT0003 administration | 48 weks
  Scale 36-Item Short From Survey (SF-36 Health Survey); from 0 (negative) to 100 (positive)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe LABRUNE, MD, PHD, Principal Investigator — APHP_Hopital Antoine BECLERE
Locations (1):
- Hopital Antoine BECLERE, Clamart, France